CLINICAL TRIAL: NCT04265560
Title: Progressive Resistance Training in Acute Spinal Cord Injury: a Pilot Randomised Controlled Trial
Brief Title: Progressive Resistance Training in Acute Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Restrictions due to COVID-19
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/WS/0149
Record Dates: First submitted 2020-01-29; First posted 2020-02-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries; Quadriplegia; Trauma, Nervous System; Paralysis; Spinal Cord Diseases
Keywords: Spinal Cord Injury; Progressive Resistance Training; Physical Therapy; Physiotherapy; Strength Training
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Trauma, Nervous System; Paralysis; Spinal Cord Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Training (Experimental): The intervention group will receive 8 weeks of Progressive Resistance Training (PRT), twice a week, in addition to usual care. An upper limb functional goal will be identified through discussion with the researcher and the participant. PRT will be individually tailored to target two muscle groups and will be chosen in order to develop strength to progress towards the participants functional goal.
  The chronic spinal cord injury exercise guideline parameters will be applied (3 sets of 8-10 repetitions, 1-2 mins rest between sets). Participants will be inducted to their PRT programme and will then independently complete the 8 week programme. During each of the following sessions, assistance for set up of equipment and/or limb position will be given by the researcher and/or the participants family, friend or carer, once they have been trained. PRT sessions will be recorded in a diary to monitor sets and repetitions completed, and intensity (visual analogue scale (VAS)).
  Interventions: Other: Progressive Resistance Training
- Usual care only (No Intervention): Participants will continue with their usual care, consistent with standard National Health Service (NHS) care in this population. Usual physiotherapy care is provided, up to 2 times per day, 4 to 5 days per week, each lasting up to 90 minutes. Physiotherapists provide a combination of group exercise and one to one function-orientated physiotherapy sessions to improve balance, general muscle strength, wheelchair and/or transfer skills.

INTERVENTIONS:
Other: Progressive Resistance Training — Progressive resistance training programme for individuals following spinal cord injury.
  Arms: Progressive Resistance Training

SUMMARY:
Muscle weakness is one of the most common and debilitating symptoms following a Spinal Cord Injury (SCI). Strength training is recommended as an effective means to increase muscular strength and improve function for individuals with long term SCI. In contrast, the strength training guidance for those with a recent (<1 year) SCI is lacking. Therefore, this study aims to investigate the feasibility of a method of upper limb strengthening - Progressive Resistance Training (PRT) and its impact upon muscle strength and function.

DETAILED DESCRIPTION:
The trial and recruitment will be conducted at the Queen Elizabeth National Spinal Injuries Unit (QENSIU), Glasgow. Individuals with tetraplegia and upper limb weakness will be randomly allocated to receive either a tailored progressive resistance training (PRT) programme alongside usual care or usual care alone.

Up to 30 participants admitted to the QENSIU will be recruited to the study. They will be randomised to the intervention or control group. The intervention group will receive 8 weeks of PRT. An upper limb functional goal will be identified through discussion with the researcher and the participant. PRT will be individually tailored to target two muscle groups which contribute to achieving this goal. For each muscle group 3 sets of 8-10 repetitions will be carried out, resistance will be applied using wrist weights, free weights or resistance bands as required. Measurements of muscle strength and function will be assessed prior to, and following the study. Outcome measures: Manual muscle testing, Handheld Dynamometry, The Spinal Cord Independence Measure, The Action Research Arm Test.

ELIGIBILITY:
Inclusion Criteria:

* Acquired non-progressive SCI - traumatic, spinal cord stroke, surgical injury
* Within 2 weeks of being identified as medically stable by the treating consultant
* Over 18 years old
* Individuals classified with complete or incomplete tetraplegia (C1-C8), graded A-D according to the American Spinal Injury Association (ASIA) scale
* Bilateral or unilateral partial paresis of at least two muscle groups of the upper limb
* Manual muscle testing grade 2-4 strength in target muscle groups
* Able to tolerate sitting upright in a wheelchair for at least 2 hours

Exclusion Criteria:

* Acute condition impairing a participant's ability to perform PRT (e.g. fracture)
* Proven or suspected neuromuscular weakness affecting the upper limbs due to another condition (e.g. stroke or Guillain-Barré syndrome)
* Unable to follow instructions in English
* Symptomatic cardiac disease
* Ventilator dependency
* Severe spasticity
* Uncontrolled autonomic dysreflexia
* Likely to be discharged before the end of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Change in muscular strength - handheld dynamometry | Baseline, 8 weeks
  Muscular strength will be quantified using handheld dynamometry, the main upper limb muscle groups will be assessed, bilaterally. Shoulder flexors, extensors, abductors, adductors, lateral rotators, and medial rotators, elbow flexors and extensors, forearm pronators and supinators, and wrist flexors and extensors will be assessed. The order of testing the muscle groups will be consistent.
  Handheld dynamometry will be conducted implementing the 'make' test. The participant will exert a maximal force against the device whilst the assessor will maintain the position of the device. Three trials will be performed for each upper limb muscle group. Prevention of muscle fatigue will be achieved by a 30-second recovery after each trial and 2 minutes rest between muscle groups. One or 2 trials will be used to familiarise participants with the testing procedure.

SECONDARY OUTCOMES:
Manual muscle testing | Baseline, 8 weeks
  Muscular strength will be quantified using manual muscle testing, the main upper limb muscle groups will be assessed, bilaterally. Shoulder flexors, extensors, abductors, adductors, lateral rotators, and medial rotators, elbow flexors and extensors, forearm pronators and supinators, and wrist flexors and extensors will be assessed. The order of testing the muscle groups will be consistent. Manual muscle testing using the Medical Research Council ordinal scale will be conducted once using standardised positions. This scale ranges from 0 to 5, 0: no palpable or visible muscle contraction, up to 5: muscle can move against gravity and maximal resistance over full range of motion.
The Spinal Cord Independence Measure (SCIM III) | Baseline, 8 weeks
  The Spinal Cord Independence Measure (SCIM III) is a measure of functional independence for individuals with SCI. It is composed of 19 items that assesses 3 domains: self-care, respiration and sphincter management and mobility. The total SCIM III scores range from 0 to 100. 0 represents total dependence, 100 represents complete independence. The blind assessor will score participants on the items for each subscale. The subscale 'self-care' exclusively relates to upper limb ability. SCIM III reflects important aspects of independence specific to the SCI population. Its use has been recommended for individuals with tetraplegia, changes within the self-care category relate to changes in upper limb function. Furthermore, it has been reported to be reliable and valid for patients with traumatic SCI.
The Action Research Arm Test (ARAT) | Baseline, 8 weeks
  Upper limb function will be assessed using The Action Research Arm Test (ARAT) following the standardised protocol outlined by Yozbatiran et al., (2008). The ARAT assesses participants ability to grasp, grip and pinch objects, and make gross motor movements. Standardised materials are required including a box with wooden blocks, alloy tubes, cups, marbles etc. Score for the ARAT ranges from 0-57 points, 57 points represents the best possible performance.
Perception of ability | 8 weeks
  At the end of the intervention period, each participant in the intervention group will be asked to rate if their functional goal has changed on a 15-point scale from -7 'a very great deal worse', to +7 'a very great deal better'.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Houliston, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No